CLINICAL TRIAL: NCT01053104
Title: Dose Adaptation of Capecitabine Using Mobile Phone Toxicity Monitoring Pilot Study of Optimal Dose Scheduling of Capecitabine for Patients With Metastatic Colorectal or Metastatic Breast Cancer
Brief Title: Dose Adaptation of Capecitabine Using Mobile Phone Toxicity Monitoring
Acronym: DATACAP
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: oxBRC (Unknown); Vodafone UK Foundation (Unknown); Centre for Statistics in Medicine (Other); Oncology Clinical Trials Office (OCTO, Oxford) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Mobile Datacap; OCTO/Oxford (Other: Trial coordinating centre)
Record Dates: First submitted 2010-01-03; First posted 2010-01-21 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Breast Cancer
Keywords: Colorectal cancer; Breast cancer; Capecitabine; Docetaxel; Mobile phone; Toxicity; Metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- capecitabine 2000mg/m2 (Colorectal): capecitabine 2000mg/m2 d 1-14, q 3 weekly and oxaliplatin 130mg/m2 d1 q 3 weekly (CAPOX)
- capecitabine 2500mg/m2 (Colorectal): capecitabine 2500mg/m2 d 1-14, q 3 weekly
- capecitabine 2000mg/m2 (Breast): capecitabine 2000mg/m2d 1-14, q 3 weekly
- docetaxel 75mg/m2 (Breast): capecitabine 2000mg/m2 d 1-14, q 3 weekly and docetaxel 75mg/m2 d1 q 3 weekly

SUMMARY:
To develop a system to manage side effects and adjust chemotherapy dose such that a patient can receive their personal maximum tolerated dose.

DETAILED DESCRIPTION:
Patients with metastatic colorectal or breast cancer will be recruited.

* Metastatic Colorectal Cancer: capecitabine alone or capecitabine + oxaliplatin for 8 3-week cycles
* Metastatic Breast Cancer: capecitabine alone or capecitabine + docetaxel for 8 3-week cycles.

All patients will be given a mobile phone onto which they will enter any side-effects experienced prior to taking capecitabine in the morning and evening. Any grade 3 or 4 symptoms will trigger an alert to a pager held by the ward-staff for immediate attention. Thus, patients' severe side-effects will be monitored in real time and the trial will allow real-time dose reductions during cycles and dose-increases at clinics. Patient experience in the trial will also be evaluated during their participation in the trial.

Patients will already be receiving the drug prior to this study and will not be administered to patients as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal or breast cancer patients commencing treatment on one of four specified regimens

For metastatic colorectal cancer:

* capecitabine 2000mg/m2 d 1-14, q 3 weekly and oxaliplatin 130mg/m2 d1 q 3 weekly (CAPOX)
* capecitabine 2500mg/m2 d 1-14, q 3 weekly

For metastatic breast cancer:

* capecitabine 2000mg/m2d 1-14, q 3 weekly
* capecitabine 2000mg/m2 d 1-14, q 3 weekly and docetaxel 75mg/m2 d1 q 3 weekly
* Age > 18 years
* Fit to start at full (100%) starting dose of all drugs
* Able and willing to use mobile phone
* Reasonable renal, liver and bone marrow function
* Absolute neutrophil count (ANC) >1.5 x 109/L
* Platelet count > 100 x 109/L
* Total bilirubin <1.5 ULN
* ALT, AST < 2.5 x ULN
* Alkaline phosphatase < 2.5 x ULN
* No obvious contra indications to capecitabine or oxaliplatin or docetaxel
* Patients must also be able to read, write and understand English.

Exclusion Criteria:

* Patients who live in an area of no Vodafone or Orange mobile phone network - - Patients participating in other cancer treatment trials
* Moderate or severe renal impairment [creatinine clearance <30ml/min (calculated according to Cockroft-Gault formula)]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Toxicities (frequency at each of grades 2, 3 and 4, over all cycles) | At the end of each cycle and at occurrence

SECONDARY OUTCOMES:
Number of inappropriate dose adaptations and self care advice messages generated ['inappropriate' defined by nurse overriding generated advice | At occurrence
Frequency of patients receiving each piece of advice from the system, including recommendations on dose and on self-treating side effects. | At occurrence
Obtain descriptive information on amount and duration of drug delivery (stage 2 only) Number of patients who, dose reduce stay at same dose dose increase Total dose delivery Chemotherapy duration | Twice daily
Obtain feedback from staff on using the system Staff recommendations for changes or improvements to the system throughout the course of the study and Semi-structured interviews | weekly for staff recommendations and one semi structured interview will take place
Test and refine mobile phone and server software systems Frequency of occurrence of technological faults (for example, problems caused by no phone reception) | At occurrence
Patient Experience EvaluationPatient experience will be evaluated as detailed in Patient Experience Evaluation | At least twice during their participation in the trial but not all patients may need to be interviewed
Evaluate safety outcomes Total number of grade 3/4 toxicities throughout the study period Degree of toxicity experienced Number of alerts, split by severity | End of each cycle and at occurrence
Dose intensity in mg/m2/week and toxicities as for stage 1 | Once at the end of the study for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Cancer Centre, Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- See also: Oncology Clinical Trials Office (OCTO) — http://www.octo-oxford.org.uk/